CLINICAL TRIAL: NCT07113886
Title: Radiographic and Histomorphometric Assessment for Guided Bone Regeneration Using a Mixture of Autogenous and Xenograft Particulate Versus Patient-Specific Sticky Bone for Horizontal Anterior Maxillary Defect (Randomized Clinical Trial)
Brief Title: Guided Bone Regeneration Using a Mixture of Autogenous and Xenograft Particulate Versus Patient-Specific Sticky Bone for Horizontal Anterior Maxillary Defect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohsen Mohamed Nasr, DR Mohamed Mohsen Mohamed Nasr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBR In Anterior Maxilla
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Sticky Bone
Keywords: ridge augmentation, horizontal bone defects, sticky bone

STUDY DESIGN:
Intervention Model Description: Interventions
  1. Preoperative preparation:
     History:
     Thorough history will be taken for all patients to identify their chief complain, medical history and dental condition. All data will be collected in the diagnostic sheet. (Appendix A)
     Clinical examination:
     • A thorough physical examination will be conducted, emphasizing the oral cavity and maxillofacial region. This includes assessing the condition of the teeth, gums, and surrounding tissues, as well as evaluating the anatomy of the maxiia .
     Consent:
     • Informed consent will be obtained from patients regarding the surgical procedure and inclusion criteria in the study
     Radiographic examination:
     • Preoperative imaging using CBCT will be performed to assess the anatomy of the maxillary bone , and the quality and quantity of bone available for grafting and to exlude the presence of any pathosis.
  2. Intra operative Surgical Procedure:
  Phase 1:
  • All surgical procedures will be performed under local Anesthesia utilizing two
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous + Xenograft particulate group. (Active Comparator)
  Interventions: Procedure: Mixture of Autogenous and Xenograft Particulates
- Patient-specific Sticky Bone group. (Experimental)
  Interventions: Procedure: Patient-Specific Sticky Bone

INTERVENTIONS:
Procedure: Mixture of Autogenous and Xenograft Particulates — This group will receive guided bone regeneration using a 1:1 mixture of autogenous bone harvested from the mandibular ramus and xenograft bone substitute (e.g., Bio-Oss). The graft material will be covered with a titanium meshes. Standard flap design, fixation, and suturing techniques will be used
  Arms: Autogenous + Xenograft particulate group.
Procedure: Patient-Specific Sticky Bone — This group will receive guided bone regeneration using patient-specific sticky bone, created by mixing autogenous bone and xenograft with autologous fibrin glue (PRF). The sticky bone graft will be molded and applied directly to the defect site, covered with a titanium meshes, and stabilized using standard surgical protocol.
  Arms: Patient-specific Sticky Bone group.

SUMMARY:
This study aims to enhance healing while minimizing invasiveness and restoring tissues to their proper structure and function by using patient specific sticky bone that will enhance the soft tissue reaction and maintain the graft volume stability and bone quality which stabilizes bone grafts, accelerates tissue healing, and reduces bone loss.

DETAILED DESCRIPTION:
II. Introduction:

6.Background and rationale:

Research question:

Does changing the bone consistency using patient specific sticky bone will enhance the soft tissue reaction and maintain the graft volume stability and bone quality if compared to the standard mix of autograft and xenograft for horizontal augmentation of anterior maxilla using guided bone regeneration? PICO Population (P): Patients with horizontal anterior maxillary defect. Intervention (I): Specific bone putty with mixture of autogenous and xenograft Comparator (C): Guided bone regeneration using mixture of autogenous and xenograft

Outcome (O):

Type of Outcome Outcome Measuring tool Unit Primary Outcome

Vertical Bone Gain

CBCT mm Secondary Outcome Horizontal Bone Gain CBCT mm Tertiary Outcome 1. Percentage of newly formed bone Histomorphometric analysis of decalcified bone sections with (H&E) stain using image analyzer computer system

Percentage (%)

2. Percentage of Mature Bone Histomorphometric analysis of decalcified bone sections with Masson's Trichome stain using Image Analyzer.computer system

Percentage (%)

Statement of the problem:

Generally, guided bone regeneration in ridge augmentation procedures often requires a collagen barrier membrane, which is intended to protect and encapsulate the graft material during the sensitive bone- remodeling phase and its integration with the native bone [26]. However, there are several drawbacks to using GBR membranes, such as the difficulty in membrane stabilization, its exorbitant cost, and rapid and unpredictable disintegration, which can result in a weakened barrier effect [27]. A study by Tony et al. proved that sticky bone does not require any collagen membrane necessity, as it alone can assist in horizontal ridge augmentation and facilitate excellent guided bone regeneration [19].

Bone augmentation is often necessary when the alveolar crest is reabsorbed and standard implants cannot be placed in a prosthetically driven position.1 Literature has validated several techniques by considering autogenous graft as the gold standard, especially for large defects. Several authors have pointed out that the outcome in large defects is better with a block graft rather than with a particulate one.2-4 Autogenous blocks need to be harvested from intraoral or extra oral sites, and this process raises the morbidity and complication rates, thereby limiting this procedure to selected patients. Moreover, the quantity of bone that can be collected from intraoral sites is limited and often it is not possible to repeat the harvesting if another area needs to be treated in the same patient.5, 6 When patients refuse intraoral harvesting or cannot stand these invasive procedures, the surgeon has several other suitable materials to use like animal-derived bone or xenograft. In the last few years, guided surgery has become an argument of discussion in modern implant treatment.11 Computer-aided oral implant surgery may offer several advantages over the traditional approach. Even regenerative surgery may have some advantages by using computer software planning. Through a computer analysis, it is possible to obtain a surgical template for implant insertion, gain information about the exact quantity of the bone defect, and fabricate a three-dimensional stereolithographic model of the patient's jaw by using a thermoplastic material that is capable of withstanding autoclave sterilization.10 The stability, effectiveness, and predictability of such a technique in horizontal defects are yet to be validated, especially when compared with the autogenous particulate mixed with demineralized bovine-bone technique.13

Rationale for conducting the research:

Sticky bone demonstrated exceptional results in various oral surgeries, effectively addressing issues such as furcation defects, bone loss, and ridge augmentation, with significant clinical and radiographic improvements. Further research is needed to explore its full potential and refine protocols for broader oral surgery and periodontics applications. "Sticky bone" is a composite biomaterial designed for bone regeneration, combining particulate bone substitutes with autologous platelet aggregates, such as PRF and concentrated growth factors (CGFs) [8]. This adaptable material conforms to various bony defects, preventing graft movement and preserving bone volume during healing, thus minimizing the need for block bone and titanium mesh. Its fibrin network captures platelets and leukocytes, releasing growth factors that accelerate bone and soft tissue regeneration without requiring biochemical additives [9]. Additionally, the fibrin interconnection prevents soft tissue ingrowth, making sticky bone suitable for treating intra-bony defects, furcation defects, ridge augmentation, and edentulous alveolar ridge defects [9]. Though studies are limited, a systematic review supports its

Review of literature:

The review's article selection process followed the PRISMA flowchart. A literature search yielded 542 relevant studies, with an additional 20 studies identified through supplementary records. After excluding 242 articles due to irrelevance, duplication, or lack of data, the screening process yielded approximately 86 articles. Of these, 48 full-text articles were assessed against eligibility criteria, resulting in the exclusion of 38 articles with explanations. Ultimately, 12 articles met the criteria and were included in the systematic review (Figure 1).

Description of Studies et al. found that sticky bone and CGF-enriched fibrin membrane improved bone quality and formation around dental implants in the narrow maxillary anterior ridge [9]. Joshi et al. showed significant gains in bone width and height with sticky bone ridge augmentation [12]. Romesh et al. reported excellent bone volume improvement using sticky bone and autologous PRF membrane for guided bone regeneration [13]. Dong-Seok et al. suggested a simplified approach to ridge augmentation with sticky bone, reducing resorption during healing [14].

In 2021, Darwish et al. evaluated socket preservation of the alveolar ridge using anorganic bovine bone and autogenous particulate bone versus sticky bone [15]. Their findings suggested increased predictability of socket preservation with sticky bone, facilitating successful implant placement. Beneytout et al. conducted a case series evaluating guided bone regeneration with PRF membrane and sticky bone graft, demonstrating its effectiveness as a supplemental approach in bone reconstruction surgery [16].

In 2022, Ghoderao et al. compared sticky bone and CGFs for intrabony osseous defects, finding superior periodontal regeneration with sticky bone [17]. Similarly, Soni et al. reported significant bone fill-in periodontal intrabony defects using sticky bone and guided tissue regeneration (GTR) membrane [18]. Tony et al. showed promising results for horizontal ridge augmentation with sticky bone, with or without a collagen membrane, leading to better horizontal bone width gain [19]. Parthasarathy et al. further supported sticky bone's efficacy in ridge augmentation through a case series [20].

In 2023, Abdelhamid et al. compared AFG to sticky bone in combination with crestal sinus lift and simultaneous implant insertion, finding favorable outcomes with sticky bone regarding implant stability and radiographic results [21]. Furthermore, Bhandari et al. presented a case report demonstrating successful periodontal regeneration of a grade III furcation defect using sticky bone alongside a PRF membrane [22].

6.b) Explanation for choice of comparators: The sticky bone can also be used in socket preservation, mainly in older patients after tooth extraction, and provides good bone quality for further implant placement. The placement of sticky bone resulted in grafted material adherence to the recipient sites without micro and macro movements, and the PRF matrix prevented early epithelial ingress onto the defect site, resulting in significant new bone gain in both horizontal and vertical dimensions [28]. Furthermore, the PRF-released growth factors, such as PDGF, epidermal growth factor (EGF), insulin-like growth factor (IGF), fibroblast growth factor (FGF), and vascular endothelial growth factor (VEGF), aid in encouraging cellular proliferation and enhance vascularity in the surgical site [28].

The sticky bone provided better bone quantity and quality in socket preservation after tooth extraction. The sticky bone was compared with anorganic bovine bone in terms of socket preservation of defective alveolar ridge and found that anorganic bovine bone showed a mean area percent of bone of 42.34%, while the sticky bone group showed 57.92% with a significant value (p < 0.05), as per Darwish et al. [15].

Management of Intra-bony Defects With Sticky Bone The sticky bone can also be packed into furcation, mainly grade III, and intra-bony defects, which showed significant tissue healing, clinical attachment gain, reduction in periodontal probing depth, and radiographic bone fill, as per Bhandari et al. [22]. These changes might have been a result of true periodontal regeneration by means of new attachment, or a long junctional epithelium between the newly regenerated tissues and the root surface. Also, sticky bone showed more promising clinical and radiographic outcomes than CGFs, as proved by Ghoderao et al. [17].

Sticky Bone in Combination With Other Biomaterials for Ridge Augmentation A study involving 28 patients found that using sticky bone and CGF combined during anterior alveolar horizontal augmentation was more effective than conventional GBR [29]. The three-dimensional architecture and mechanical characteristics of three combinations of autologous platelet liquid (APL), blood, or physiological water, and composite bovine graft, were assessed in a previously conducted in vitro study [30]. The mechanical resistance increased by 875% when APL and bone graft were combined, according to the results. With the creation of a composite sticky graft block and enhanced clinical strategies, this combination of biomaterials could improve the maxillary bone defects treatments. The clinical outcomes of guided bone regeneration using the bone-shell technique and sticky bone in horizontal ridge augmentation were compared in a prior retrospective study. Eighty patients had the bone-shell technique and sticky bone, and CBCT was used to measure the ridge widths before and six months after surgery. Records were maintained on implant survival rate and post-operative complications. The two groups' results were not different significantly, and there was no record of implant failure. Clinical results were comparable for bone-shell technique and sticky bone. Despite the initial complications and patient dropouts, the remaining participants showed consistent improvement in ridge width without significant differences between the test and control groups. Additionally, all implants remained successful over the follow-up period, indicating a positive long-term outcome [31].

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders requiring implants placement in anterior maxilla with horizontal bone defect.
* Patients of age older than 20 years old.
* Patients with adequate Inter-arch space.
* Patients who were willing and fully capable to comply with the study protocol.

Exclusion Criteria:

* Heavy smokers (> than 10 cigarettes a day)
* Patients with parafunctional habits
* Patients with uncontrolled systemic diseases.
* Patients with poor oral hygiene
* Patients with mental instabilities or psychic patient

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic and Histomorphometric Assessment for Guided Bone Regeneration using a Mixture of Autogenous and Xenograft Particulate Versus Patient-Specific Sticky Bone for Horizontal Anterior Maxillary Defect (Randomized Clinical Trial) | Baseline (preoperative), 6 months postoperative for radiographic evaluation; 6 months postoperative for histomorphometric biopsy assessment at re-entry.
Radiographic and Histomorphometric Assessment for Guided Bone Regeneration using a Mixture of Autogenous and Xenograft Particulate Versus Patient-Specific Sticky Bone for Horizontal Anterior Maxillary Defect (Randomized Clinical Trial) | Baseline (preoperative), 6 months postoperative for radiographic evaluation; 6 months postoperative for histomorphometric biopsy assessment at re-entry.
  Radiographic outcomes will include CBCT-based measurements of horizontal ridge width and bone volume gain at the grafted sites. Histomorphometric evaluation will be performed using biopsies collected at re-entry to assess new bone formation, residual graft particles, and connective tissue. Comparisons will be made between autogenous/xenograft particulate grafts and patient-specific sticky bone in terms of bone regeneration effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ass. Prof. Dr. Mohamed Mounir Mounir Associate professor of Oral and Maxillofacial Surgery, Associate professor, Principal Investigator — Oral & Maxillofacial Surgery Faculty of Dentistry - Cairo University
Locations (1):
- Oral & Maxillofacial Surgery Faculty of Dentistry - Cairo University, Cairo, Egypt